CLINICAL TRIAL: NCT01597661
Title: Bupropion and Cardiac Birth Defects (Slone Epidemiology Center)
Brief Title: Bupropion & Cardio Birth Defect (Slone)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115433; WEUSKOP5344 (Other: GSK); EPI40662 (Other: GSK)
Record Dates: First submitted 2012-02-02; First posted 2012-05-14 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Depressive Disorder
Keywords: first trimester; left outflow tract obstruction; Bupropion; cardiovascular malformation; antidepressants; pregnancy; cardiovascular defect; congenital malformation
MeSH Terms: conditions — Depressive Disorder; Congenital Abnormalities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Malformed and population-based sample of non-malformed infants: Infants with any of a wide range of malformations are identified at tertiary care and birth hospitals in four study centers (Boston, Philadelphia, Toronto, San Diego) using approaches that include reviewing lists of discharge diagnoses available in medical records; contacting newborn nursery and/or labor and delivery rooms; reviewing admission/discharge lists; and reviewing clinic and surgical logs. A population-based random sample of non-malformed newborns in Massachusetts is also included. Information gathered on each subject includes name, address, telephone number, diagnostic information, and date of birth.
  Interventions: Drug: Exposure to any bupropion during the first trimester; Drug: Exposure to bupropion alone during the first trimester; Other: Referent group: no exposure to any anti-depressant or anti-smoking drug during pregnancy

INTERVENTIONS:
Drug: Exposure to any bupropion during the first trimester — The primary exposure group will be: any exposure to bupropion during the time period from 28 days prior to the last menstrual period through the fourth lunar month. The use of bupropion in combination with other anti-depressants, exposure to SSRI anti-depressants, and exposure to non-SSRI anti-depressants, including tricyclic anti-depressants, during this time period will be explored.
  Mothers of identified infants are contacted within 6 months of delivery and invited to participate in the study by completing a telephone interview, conducted by trained study nurses. The interview addresses demographic, reproductive, and medical factors; medication and vitamin use; cigarette smoking, alcohol, and caffeine consumption, occupational exposures, and dietary intake. Exposure information is obtained directly from the mother in response to questions that focus both on indications for medication use and on medications themselves.
Drug: Exposure to bupropion alone during the first trimester — The secondary exposure group will be: bupropion exposure alone during the time period from 28 days prior to the last menstrual period through the fourth lunar month.
  Mothers of identified infants are contacted within 6 months of delivery and invited to participate in the study by completing a telephone interview, conducted by trained study nurses. The interview addresses demographic, reproductive, and medical factors; medication and vitamin use; cigarette smoking, alcohol, and caffeine consumption, occupational exposures, and dietary intake. Exposure information is obtained directly from the mother in response to questions that focus both on indications for medication use and on medications themselves.
Other: Referent group: no exposure to any anti-depressant or anti-smoking drug during pregnancy — The referent group will be defined as no exposure to any anti-depressant or anti-smoking drug at any time from 28 days prior to the last menstrual period through the end of pregnancy.
  Mothers of identified infants are contacted within 6 months of delivery and invited to participate in the study by completing a telephone interview, conducted by trained study nurses. The interview addresses demographic, reproductive, and medical factors; medication and vitamin use; cigarette smoking, alcohol, and caffeine consumption, occupational exposures, and dietary intake. Exposure information is obtained directly from the mother in response to questions that focus both on indications for medication use and on medications themselves.

SUMMARY:
Bupropion is a unique drug that is used both to treat depression and as an aid in smoking cessation. In 2008, the final report from the Bupropion pregnancy registry described 24 congenital malformations among the 675 women exposed to bupropion in the first trimester of pregnancy. Of these, 9 had congenital heart disease of varying severity, including a number of infants with ventricular septal defects (VSDs); of note, 2 of these 9 had coarctation of the aorta. More recently, Alwan et al, in an analysis of data from the Centers for Disease Control and Prevention's case-control National Birth Defects Prevention Study, reported an increased risk of left outflow tract heart defects, a subgroup of cardiac malformations that includes coarctation of the aorta and hypoplastic left heart syndrome.

Data from the Slone Epidemiology Center Birth Defects Study will be used to test these observations. The outcomes of primary interest will include those hypothesized to be associated with bupropion in recent studies: left outflow tract defects considered as a group. Coarctation of the aorta and hypoplastic left heart syndrome will also be examined separately. All infants with congenital heart defects are further classified into subgroups that are embryologically meaningful, including left outflow tract defects. In secondary analyses, other heart defect classes for which there are adequate numbers of cases will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with congenital heart defects who are born within the catchment areas of the 4 study centers
* A sample of nonmalformed infants born at participating hospitals
* Subjects who were interviewed in 1992 or later
* Women who complete the study interview within 6 months of the infant's birth

Exclusion Criteria:

* Infants with chromosomal anomalies

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The primary focus of the Slone Epidemiology Center Birth Defects Study (BDS) case-control surveillance is to identify the risks and safety of marketed drugs taken by pregnant women. Infants with any of a wide range of malformations are identified at tertiary care and birth hospitals in four study centers (Boston, Philadelphia, Toronto, San Diego) using approaches that include reviewing lists of discharge diagnoses available in medical records; contacting newborn nursery and/or labor and delivery rooms; reviewing admission/discharge lists; and reviewing clinic and surgical logs. Information gathered on each subject includes name, address, telephone number, diagnostic information, and date of birth. Beginning in 1992, the BDS also included mothers of non-malformed infants: initially these infants were identified exclusively at study hospitals, but in 1998, they expanded their normal newborn capability by obtaining a population-based random sample of newborns in Massachusetts.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2011-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Diagnosis of left outflow tract defects | Within 6 months of delivery
Diagnosis of coarctation of the aorta | Within 6 months of delivery
Diagnosis of hypoplastic left heart syndrome | Within 6 months of delivery

SECONDARY OUTCOMES:
Diagnosis of other congenital heart defects | Within 6 months of delivery

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline